CLINICAL TRIAL: NCT02569021
Title: Battery-preserving Stimulation Patterns to Improve Symptoms in Parkinson's Disease and Essential Tremor
Brief Title: Battery-preserving Stimulation Patterns for Deep Brain Stimulation
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501030
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Parkinsons Disease; Essential Tremor
Keywords: Parkinsons Disease; Essential Tremor; DBS; Depp Brain Stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Biphasic DBS stimulations: Subjects in this group will have Biphasic DBS stimulation setting performed, Unified Parkinson's Disease Rating Scale (UPDRS), Tremor Rating Scale (TRS), kinesia accelerometer assessment, Trigno wireless system (EMG) assessment and GaitRite walking assessment performed.
  Interventions: Device: Biphasic DBS stimulation; Other: Unified Parkinson's Disease Rating Scale; Other: Tremor Rating Scale; Device: Kinesia accelerometer; Device: Trigno wireless system; Other: GaitRite walking assessment.

INTERVENTIONS:
Device: Biphasic DBS stimulation — The following protocol will be followed for each subject. In between, baseline and novel stimulation settings there will be a 30-minute washout period with DBS in the off state.
  1. Current best/optimized DBS setting (considered "baseline")
  2. DBS off for 30 minutes as a washout period
  3. Biphasic pulse stimulation mode (assessment at 0.5hr)
  4. Biphasic pulse stimulation mode (assessment at 1hr)
  5. Biphasic pulse stimulation mode (assessment at 2hr)
  6. Biphasic pulse stimulation mode (assessment at 3hr)
Other: Unified Parkinson's Disease Rating Scale — UPDRS is used by neurologists to rate the motor impairment of people with Parkinson's Disease.
  Other Names: UPDRS
Other: Tremor Rating Scale — TRS is used by neurologists to rate the severity of a tremor.
  Other Names: TRS
Device: Kinesia accelerometer — The kinesia accelerometer is used to analyze the tremor and slowness (bradykinesia) of the participants.
Device: Trigno wireless system — The Trigno system measure muscle contractions.
Other: GaitRite walking assessment. — GaitRite records a patients gait pattern.

SUMMARY:
The purpose of this research study is to test effectiveness of different deep brain stimulation (DBS) stimulation patterns on symptoms that may also improve the life of the battery. If these patterns are effective, the implanted batteries will be drained more slowly and last longer than currently expected. An increase in battery life may reduce the number of surgeries needed to replace them.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an effective surgical therapy for medication-refractory symptoms of Parkinson's disease, tremor, and dystonia. Patients implanted with DBS experience a significant improvement of their symptoms with relatively low risk of intolerable side effects. Implanted patients must undergo repeat surgeries to replace the Implantable Pulse Generators/batteries (IPG) approximately every 2 to 5 years. The DBS program (at the University of Florida) has studied battery consumption and has been interested in potential strategies to extend the life of the IPG to reduce the need for frequent battery replacement surgeries, while improving symptom-relief, patient satisfaction, and the potential associated financial burdens.

The research study will evaluate the effects of novel stimulation patterns on tremor, bradykinesia, rigidity and gait in Parkinson's disease and essential tremor patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease or Essential Tremor by strict criteria
* Deep brain stimulation (DBS) already implanted
* Optimized Deep brain stimulation (DBS) settings (or at least 4 months of DBS programming)

Exclusion Criteria:

* Other neurological diagnoses (co-existent Alzheimer's or ALS)
* No Deep brain stimulation (DBS)
* less than 4 Deep brain stimulation (DBS) programming

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during routine DBS programming sessions at the University of Florida, Center for Movement Disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of novel stimulation patterns by the Unified Parkinson's Disease Rating Scale | Baseline to Day 1
  The Unified Parkinson's Disease Rating Scale (UPDRS) is used by neurologists to rate the motor impairment of people with Parkinson's Disease. The rater obtains the score by observation and questioning the participant. Higher scores represent greater impairment and scores range from 0-108. The subject will be videotaped and two raters blinded to conditions will score the UPDRS.
Evaluate the efficacy of novel stimulation patterns by the Tremor Rating Scale | Baseline to Day 1
  Tremor Rating Scale (TRS), consists of 11 items that evaluate tremor in the head, arms, and legs. The rater assigns a score of 0 to 4 for each item, in ascending order of severity. The subjet will be videotaped and two raters blinded to conditions will score the TRS.
Kinesia accelerometer to measure motor dysfunction | Baseline to Day 1
  The Kinesia system includes a unit worn by the subject and software that is used to collect, manage, and analyze data. The system measures three-dimensional motion using three orthogonal accelerometers and three orthogonal gyroscopes located in the sensor module.The digital data is received by the Receiver connected to a computer and processed by the Kinesia software package.
Trigno wireless system to measure motor dysfunction | Baseline to Day 1
  This system has sensors with a multi-function design and therefore along with recording of surface EMG signal, it allows Triaxial Accelerometry. This wireless EMG machine will measure muscle contractions.
GaitRite walking assessment. | Baseline to Day 1
  The GaitRite is an automated floor that when the subjects walk on the floor it records the gait pattern.

SECONDARY OUTCOMES:
Battery Consumption compared between pre and post settings | Baseline to Day 1
  Battery consumption will be calculated and compared between the new settings and subjects' baseline settings. The Medtronic battery estimator helpline will be used to calculate battery life, as well as the University of Florida calculator.

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Okun, M.D., Principal Investigator — University of Florida
Locations (1):
- Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States